CLINICAL TRIAL: NCT06239363
Title: Nutritional Sources of Salicylates and Disorders of Placental Angiogenesis in Preeclampsia
Brief Title: Dietary Salicylates and Preeclampsia
Acronym: PreSal
Status: Recruiting | Type: Observational
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Joanna Suliburska, professor, Poznan University of Life Sciences
Other Study IDs: 34/2023
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy Disease; Preeclampsia; Diet Habit
Keywords: pregnancy; preeclampsia; angiogenesis; salicylates
MeSH Terms: conditions — Pre-Eclampsia; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preeclampsia (PE) is an important pregnancy complication and cause of maternal and perinatal mortality and morbidity. The underlying etiology and pathophysiology of preeclampsia is incompletely understood but it involves dysfunctional cytotrophoblastic invasion, placental ischemia, and release of inflammatory and endothelial mediators. Placenta dysfunction in PE is related to angiogenic balance. Currently, therapeutic options for the prevention and treatment of PE are limited. It is known that the risk of PE is reduced by low-dose aspirin. Therefore, the influence of salicylates on the development of PE seems to need to be investigated. This project plans to examine the preventive effects of food sources of salicylic acid and compare their effects with aspirin. Therefore, the aim of the present study is thus answer the following questions. whether the maternal dietary intake of salicylates is related to placental angiogenesis; 2. whether naturally occurring salicylates have the same effects on preeclampsia development and placental angiogenesis as aspirin. To answer these questions we plan to carry out a human study with pregnant women.

Due to the above the planned research aims to determine the association between maternal dietary intake of salicylates and placental angiogenesis and the risk of preeclampsia development.

Although PE remains an incurable disease, the results of this project will enable the development of dietary recommendations for the prevention and treatment of preeclampsia. Moreover, the results of this study may be useful in lowering the cost of maternal and fetal complications from preeclampsia and the cost of their hospitalization.

DETAILED DESCRIPTION:
Preeclampsia (PE) is one of the most important complications in pregnancy worldwide and is responsible for over 70,000 maternal deaths each year around the world. Babies born to women with PE often suffer from intrauterine growth restriction and preterm birth along with increased fetal pro-inflammatory profiles which require a long and costly hospitalization. PE results in placental dysfunction and it is now accepted that PE is a placental disease. Placenta dysfunction in PE is related to impaired angiogenic balance. Currently, therapeutic options for the prevention and treatment of PE are limited. It is known that the risk of PE is reduced by low-dose aspirin.

Therefore, the influence of salicylates on the development of PE seems to need to be investigated.

This project plans to examine the preventive effect of natural salicylates and compare their effects with aspirin. Therefore, the aim of the present study thus answer the following questions. whether the maternal dietary intake of natural salicylates is related to placental angiogenesis; 2. whether naturally occurring salicylates have the same effects on preeclampsia development and placental angiogenesis as aspirin.

The study will aim to determine the association between maternal dietary intake of salicylates and placental angiogenesis and the risk of preeclampsia development.

The study will be carried out in around 500 pregnant women (healthy and with PE) aged 18-45 years.

Daily food intake will be determined based on the FFQ questionnaire and dietary intake interviews. The amount of salicylic acid and total salicylates in the daily diet will be processed and evaluated.

Blood samples were collected from a maternal vein at the time of delivery. In plasma, it will be assayed salicylates, salicylic acid, TNFα, and hsCRP concentrations. Biomarkers of angiogenesis will be assayed in plasma: concentration of VEGF, PLGF, and sFLT1.

The placentas will be collected after delivery. Biomarkers of angiogenesis will be assayed in the placenta: concentration of VEGF, PLGF, and sFLT1. In the placenta, it will be measured mRNA and proteins of STOX 1. The vascularization process will be evaluated in the placenta.

Women will collect 24-hour urine. Salicylates and salicylic acid will be assayed in urine.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* healthy women with no previous adverse medical history and women with diagnosed preeclampsia
* singleton pregnancy
* people who have the full ability to give informed consent.

Exclusion Criteria:

* pregnancies with detectable fetal defects, chromosomal abnormalities, genetic syndromes
* infections
* history of chronic hypertension, metabolic disorder before or during pregnancy, or the presence of high-risk factors such as heart diseases, diabetes, and renal diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The study will be carried out in around 500 pregnant women (healthy and with preeclampsia) aged 18-45 years.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
daily intake using 24-hour Dietary Recall | 3 years
  evaluation of daily intake of nutrients (carbohydrate, fat, protein, vitamins, minerals, energy)
salicylates | 3 years
  measure in plasma and urine
angiogenesis biomarker: sFLT1 | 3 years
  measure in plasma and placenta
angiogenesis biomarker: VEGF | 3 years
  measure in plasma and placenta
angiogenesis biomarker: PLGF | 3 years
  measure in plasma and placenta
STOX-1 protein | 3 years
  measure in placenta
inflammatory biomarker: TNFα | 3 years
  measure in plasma
inflammatory biomarker: hsCRP | 3 years
  measure in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland